CLINICAL TRIAL: NCT02474797
Title: Assessment of Diaphragmatic Function by Ultrasonographic Measure of Diaphragmatic Thickening in Severe Sepsis or Septic Shock Patients Hospitalized in ICU: Diaphragmatic Dysfunction Frequency, Prognosis Values and Associated Factors
Brief Title: Ultrasound Diaphragmatic Thickening to Monitor Its Dysfunction in Patients With Sepsis
Acronym: US-Diamonds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2014-A01942-45
Record Dates: First submitted 2015-06-03; First posted 2015-06-18 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Sepsis; Disease of Diaphragm; Defect of Diaphragm; Intensive Care Neuropathy
Keywords: Ultrasonography; Diaphragm; Lung ultrasound; Sepsis; Critical care; Chest physiotherapy
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diaphragmatic ultrasonography in septic patient (Experimental): Diaphragmatic Thickening Fraction
  Interventions: Device: Diaphragmatic ultrasonography

INTERVENTIONS:
Device: Diaphragmatic ultrasonography — Daily Measure of Diaphragmatic Thickening Fraction (DTF) will be performed by a trained physiotherapist. Physiotherapist (A. LE NEINDRE). The patient will be then instructed to perform breathing to total lung capacity and then to exhale to residual volume, when it is possible (awaken patient). Awakening status will be recorded. Mechanically ventilated patients will be evaluated in Pressure Support (PS) mode (during daily PS mode research for patients with Controlled Ventilation), with the lower PS level tolerated. PS level will be recorded.
  Thickening fraction (TF) measure is performed in B-mode using the following formula: TF (%) = [(end-inspiration thickness - end-expiration thickness)/(end-expiration thickness) x 100]. Diaphragmatic dysfunction is defined like a DTF < 20% (7).
  Other Names: Diaphragmatic sonography

SUMMARY:
Diaphragmatic dysfunction is associated with sepsis severity and pejorative prognosis. Aim of this study is to assess diaphragmatic function with the Diaphragmatic Thickening Fraction (DTF) ultrasound measure in patients with severe sepsis or septic shock, mechanically ventilated or not, hospitalized in ICU in order to determinate diaphragmatic dysfunction frequency, its prognosis value and its associated factors.

This is a prospective pilot study in a 14-bed medical and surgical ICU including 50 consecutive patients with severe sepsis or septic shock. The expected duration of study is 18 months.

DTF is measured each day as follow: the probe is placed in an intercostal space between mid axillary line and anterior axillary line, 0.5cm to 2 centimeters below the costodiaphragmatic sinus. DTF measure is performed in B-mode using the following formula: TF (%) = [(end-inspiration thickness - end-expiration thickness)/(end-expiration thickness) x 100]. A DTF < 20% indicates a diaphragmatic dysfunction.

The investigators will collect potential factors for which DTF Ultrasound Measure could have a prognosis value (intubation, successful or failed weaning from mechanical ventilation), potential risk factors (age, sex, tobacco, alcohol etc.) and potentials associated factors.

The investigators expect measure of DTF allows identifying patient with severe sepsis or septic shock with diaphragmatic dysfunction. It would also estimate diaphragmatic dysfunction frequency with ultrasound measure and warranting its use routinely at the bedside. The investigators expect that DTF helps to characterize degree of severity of septic patient and can be a new index able to predict intubation in this population.

DETAILED DESCRIPTION:
Rational Severe sepsis and septic shock represent the first cause of death in ICU (42% to 60% mortality rate). Sepsis is defined by alteration of cellular function, immune dysregulation, coagulation and metabolism disorders, following the Systemic Inflammatory Response Syndrome (SIRS).

Among different affected organs, skeletal muscle is highlighted. Proteolysis increasing, proteosynthesis decreasing and mitochondrial dysfunction lead to an overall muscular cells alteration (sarcolemma, sarcoplasmic reticulum and contractile proteins). These mechanisms induce a reduction of skeletal muscle mass and skeletal muscle-specific force generation. Diaphragm could be the first muscle affected during sepsis (1). Sepsis is the primary risk factor for diaphragmatic dysfunction. Diaphragm could be considered as an organ altered by sepsis (2). Diaphragmatic dysfunction is associated with sepsis severity and pejorative prognosis. Its assessment becomes an important issue in order to evaluate the patient severity status, to monitor diaphragm recovery and adjust treatment.

One study evaluated diaphragmatic function with Magnetic Phrenic Nerve Stimulation in mechanically ventilated patients (3) and one with Needle Electromyography of diaphragm in patients with prolonged weaning from mechanical ventilation (4). But any study assessed diaphragmatic function with ultrasound measure of Diaphragmatic Thickening Fraction in patients with severe sepsis or septic shock, mechanically ventilated or not.

Ultrasonography is noninvasive, ionization free, feasible rapidly at the bedside and thus can be regularly used in diaphragm assessment (5). The diaphragmatic thickening fraction (DTF) at the zone of apposition (6) allows to assess thickening capacity of diaphragm during inspiration so its contraction capacity. It is an accurate and reproducible outcome measure for diaphragmatic dysfunction assessment. A DTF < 20% indicates a diaphragmatic dysfunction (7).

We hypothesize that acute diaphragmatic abnormalities are present in ICU septic patient and it can be a prognosis factor of patient severity.

Aim of this study is to assess diaphragmatic function with the DTF ultrasound measure in patients with severe sepsis or septic shock, mechanically ventilated or not, hospitalized in ICU in order to determinate diaphragmatic dysfunction frequency, its prognosis value and its associated factors.

Objectives Primary To estimate diaphragmatic dysfunction frequency with measure of Ultrasound DTF in ICU septic patients.

Secondary:

* To determine if DTF is a predictor of intubation;
* To determine if DTF is a predictor of successful weaning from mechanical ventilation in subgroup of mechanically ventilated patients;
* To monitor changes of DTF during ICU hospitalization;
* To determine risk factors of diaphragmatic dysfunction;
* To determine associated factors of diaphragmatic dysfunction.

Methods Design This is a prospective study in a 14-bed medical and surgical ICU including 50 consecutive patients with severe sepsis or septic shock.

Data collections Demographic data, antecedents, severity score, organ dysfunction-related variables, physiologic data, presence of sepsis, presence of mechanical ventilation and medications will be prospectively recorded on inclusion (ICU admission for severe sepsis/septic shock or severe sepsis/septic shock occurring during ICU hospitalization). Ultrasound DTF, severity score, organ dysfunction-related variables, physiologic data, presence of septic shock, medications, presence of mechanical ventilation will be prospectively recorded each days of ICU hospitalization. Duration of mechanical ventilation, number of failed extubation, decision to perform tracheostomy, ICU and Hospital stay, ICU and Hospital mortality will be also recorded.

Recruitment Patients will be recruited in a 14-bed medical and surgical ICU when they present inclusion criteria.

All patients or their relatives will provide written consent to participate.

Diaphragm thickening assessment All patients will be evaluated in a semi-recumbent position. Ultrasound will be performed using an ultrasound system equipped with a 10 megahertz linear probe.

Daily Measure of Diaphragmatic Thickening Fraction (DTF) will be performed by a trained physiotherapist. Physiotherapist (A. LE NEINDRE) was trained during six months for this measure by a well-trained Physician.

DTF is measured each day as follow (7): the probe is placed in an intercostal space between mid axillary line and anterior axillary line, 0.5cm to 2 centimeters below the costodiaphragmatic sinus. With B-mode the diaphragm is observed like a structure made of three distinct layers: a nonechogenic central layer bordered by two echogenic layers: pleural line (internal layer) and peritoneum (external layer).

The patient will be then instructed to perform breathing to total lung capacity and then to exhale to residual volume, when it is possible (awake patient). Awakening status will be recorded. Mechanically ventilated patients will be evaluated in Pressure Support (PS) mode (during daily PS mode research for patients with Controlled Ventilation), with the lower PS level tolerated. PS level will be recorded.

DTF measure is performed in B-mode using the following formula: TF (%) = [(end-inspiration thickness - end-expiration thickness)/(end-expiration thickness) x 100]. Three consecutive measures will be performed. Video files will be recorded and DTF will be estimated independently by a second trained operator (Dr F. PHILIPPART), unaware of patient conditions. The better value of these three measures will be retained. Diaphragmatic dysfunction is defined like a DTF < 20% (7).

Assessment of DTF reproducibility Twenty recordings (from twenty separate patients) will be randomly selected from the study to assess analyzer reproducibility. The same sets of recording will be analyzed twice by the same Ultrasound Performer (A. LE NEINDRE) to assess intra-analyzer reproducibility and separately by two different Ultrasound Performers (A. LE NEINDRE and F. PHILIPPART) to assess inter-analyzer reproducibility.

Statistical Analysis Diaphragmatic dysfunction frequency is defined by proportion of patient with DTF<20%. It will be expressed as a percentage with 95% Confidence Interval.

Receiver Operating Characteristic (ROC) curve analysis will be performed to assess DTF ability to discriminate between patients who will be intubated and those who will be not. ROC curve analysis will be also used to discriminate mechanically ventilated patients who will fail to wean and those who will success.

DTF will be analyzed as a continuous variable and univariate linear regression models will be used to identify factors associated with higher or lower DTF values. Multivariate analysis will be performed using a forward logistic regression process taking into account all potential associated factors for diaphragm dysfunction.

Each potential risk factor for diaphragm dysfunction (DTF < 20%) will be evaluated in a univariate model (Student t or Mann-Whitney U test for continuous variables depending on distribution; chi-square test or Fisher exact test for categorical variables depending on size), and multivariate analysis will be performed. For all comparisons, a P value less than or equal to 0.05 will be considered statistically significant.

Impact of Diaphragmatic dysfunction on ICU and hospital mortalities, institution of mechanical ventilation, failed weaning form mechanical ventilation, tracheostomy rate will be assessed.

Impact of Diaphragmatic dysfunction on ICU and hospital mortalities will be evaluated using Kaplan-Meier survival function estimates.

Expected results We expect measure of DTF allows identifying patient with severe sepsis or septic shock with diaphragmatic dysfunction. It would also estimate diaphragmatic dysfunction frequency with ultrasound measure and warranting its use routinely at the bedside. We expect that DTF helps to characterize degree of severity of septic patient and can be a new index able to predict intubation in this population. As previous studies showed in other populations, DTF could predict success of extubation in mechanically ventilated septic population. It would be another tool to monitor evolution of organ failure. A second study will be conduct in order to evaluate a new strategy to manage septic patient at risk of diaphragmatic dysfunction (Inspiratory Muscle Training) and the use of DTF as a predictive index of intubation.

Organization of the project Number of Participants This is a pilot study aiming to establish diaphragmatic dysfunction frequency, prognosis and associated factors in patients with severe sepsis or septic shock. We wish a 18 months maximal duration of study. Considering the recruiting capacity of our ICU and our previous studies for this population we will include 50 consecutive patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in our Medical/Surgical ICU;
* Severe sepsis of septic shock (2001 International Sepsis Definition Conference);
* Age > 18 years;
* Patient consent.

Exclusion Criteria:

* Preexisting neuromuscular disorders;
* Recent cardiac or thoracic surgery;
* Use of neuromuscular blocking agent within the 24h preceding the first diaphragm assessment;
* Known preexisting diaphragmatic disorders;
* Cervical spine injury;
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic Dysfunction with DTF Ultrasound measure | Participants will be followed for the duration of ICU stay, an expected average of 10 days
  Diaphragmatic dysfunction is defined by DTF < 20%. Frequency of diaphragmatic dysfunction is measured by the ratio of: number of patient with DTF < 20% during ICU hospitalization on total number of patients included.

SECONDARY OUTCOMES:
Collection of potential factors for which DTF Ultrasound Measure could have a prognosis value: intubation, successful or failed weaning from mechanical ventilation | Participants will be followed for the duration of ICU stay, an expected average of 10 days
Collection of potential risk factors: age, sex, tobacco, alcohol, cirrhosis, diabetes mellitus | At baseline
Collection of potentials associated factors: medication (hypnotics, opioids, steroids, catecholamines), mechanical ventilation, presence of a septic shock, severity score (SOFA), ICU and Hospital Length of stay, ICU and Hospital mortality | Participants will be followed for the duration of ICU stay, an expected average of 10 days
Change in Diaphragmatic Thickening Fraction with DTF Ultrasound measure | Participants will be followed for the duration of ICU stay, an expected average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Aymeric Le Neindre, PT, MSc, Principal Investigator — Fondation Hôpital Saint-Joseph; François Philippart, MD, PhD, Principal Investigator — Fondation Hôpital Saint-Joseph; Benoît Misset, MD, PhD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Jung B, Nougaret S, Conseil M, Coisel Y, Futier E, Chanques G, Molinari N, Lacampagne A, Matecki S, Jaber S. Sepsis is associated with a preferential diaphragmatic atrophy: a critically ill patient study using tridimensional computed tomography. Anesthesiology. 2014 May;120(5):1182-91. doi: 10.1097/ALN.0000000000000201. PMID 24608360
- [Background] Supinski GS, Callahan LA. Diaphragm weakness in mechanically ventilated critically ill patients. Crit Care. 2013 Jun 20;17(3):R120. doi: 10.1186/cc12792. PMID 23786764
- [Background] Demoule A, Jung B, Prodanovic H, Molinari N, Chanques G, Coirault C, Matecki S, Duguet A, Similowski T, Jaber S. Diaphragm dysfunction on admission to the intensive care unit. Prevalence, risk factors, and prognostic impact-a prospective study. Am J Respir Crit Care Med. 2013 Jul 15;188(2):213-9. doi: 10.1164/rccm.201209-1668OC. PMID 23641946
- [Background] Santos PD, Teixeira C, Savi A, Maccari JG, Neres FS, Machado AS, de Oliveira RP, Ribeiro M, Rotta FT. The critical illness polyneuropathy in septic patients with prolonged weaning from mechanical ventilation: is the diaphragm also affected? A pilot study. Respir Care. 2012 Oct;57(10):1594-601. doi: 10.4187/respcare.01396. Epub 2012 Mar 13. PMID 22417531
- [Background] Bouhemad B, Zhang M, Lu Q, Rouby JJ. Clinical review: Bedside lung ultrasound in critical care practice. Crit Care. 2007;11(1):205. doi: 10.1186/cc5668. PMID 17316468
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Summerhill EM, El-Sameed YA, Glidden TJ, McCool FD. Monitoring recovery from diaphragm paralysis with ultrasound. Chest. 2008 Mar;133(3):737-43. doi: 10.1378/chest.07-2200. Epub 2008 Jan 15. PMID 18198248